CLINICAL TRIAL: NCT04426812
Title: Measuring Chronic Pain Impact
Brief Title: Measuring Chronic Pain Impact: Measurement Enhancement for Chronic Pain
Status: Completed | Type: Observational
Sponsor: RAND (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: RHINO ID 2019-0651
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MTurk sample: Data collected from a sample of participants in an online convenience platform called MTurk who self-identify as having chronic pain.
  Interventions: Other: No intervention; just data collection
- KnowledgePanel: Data collected from a sample of panel members in an online representative panel called KnowledgePanel who self-identify as having chronic pain.
  Interventions: Other: No intervention; just data collection

INTERVENTIONS:
Other: No intervention; just data collection — No intervention; just data collection

SUMMARY:
Many complementary and integrative health approaches have been shown to be effective for chronic pain and included in guidelines. This evidence of effectiveness is built on hundreds of studies representing millions of research dollars, and the ability to analyze and better compare results across these studies is essential to obtain the full value of this investment. However, useful across-study comparisons which would allow better understanding and targeting of these interventions are hampered by at least two challenges: the lack of common outcome measures and the inability to meaningfully stratify or classify patients.

The first two Aims of this study each address one of these two challenges. The last Aim takes advantage of this study to further test the viability of MTurk as a data collection platform.

Specific Aim 1 addresses the lack of common outcome measures. This Aim is to develop and evaluate links or crosswalks between the PROMIS-29 and other common (legacy) measures used for chronic pain so that the results of studies using different measures can be compared. Our hypothesis here is that we will be able to create some sort of linkage between PROMIS and legacy measures that will allow for each pair estimates of one to be made from the other.

Specific Aim 2 addresses the inability to meaningfully stratify or subclassify chronic pain patients. This Aim is to evaluate and refine the chronic pain impact stratification scheme (ISS) proposes by the NIH Research Task Force on chronic low back pain, which is based on 9 PROMIS-29 items. Our hypothesis here is that the ISS can be refined so that it can identify subgroups of chronic pain patients with different levels of morbidity and different needs for treatment.

Specific Aim 3 addresses the potential for more efficient data collection using the MTurk platform. This Aim is to evaluate MTurk as a cost- and time-efficient method to collect quality data on individuals with chronic pain. Our hypothesis here is that we find that MTurk produces data of sufficient quality to be of use to future research projects.

DETAILED DESCRIPTION:
While there is an extensive literature on the effectiveness of pharmaceutical and nonpharmacologic interventions for chronic low back pain (CLBP), it is challenging to synthesize the findings because of differences in the CLBP samples and in the outcome measures used. The NIH Research Task Force (RTF) on CLBP noted that these differences make it "difficult to compare epidemiologic data and studies of similar or competing interventions, replicate findings, pool data from multiple studies, resolve conflicting conclusions, develop multidisciplinary consensus, or even achieve consensus within a discipline regarding interpretation of findings." To this list we would add that these differences also prevent the use of the results to answer questions such as 'Which therapies work best? And for whom?' This project tackles two things that are needed to address these differences and allow for better cross-study comparisons: we will develop empirical links between different outcome measures to allow their expression in similar units (Aim 1), and we will refine the RTF's proposed stratification (subgrouping) of patients by the impact of their CLBP (Aim 2).

To address the first challenge, in Aim 1 this study will develop and evaluate crosswalks or links between components of the 29-item Patient-Reported Outcomes Measurement Information System (PROMIS®) short form (PROMIS-29) and common legacy measures used for chronic pain. The purpose of these crosswalks or links is to allow researchers who measured outcomes using one instrument to estimate what the outcome would be if it had been measured using the other instrument. In particular, we will create crosswalks/links for the two most commonly used instruments used to measure outcomes for CLBP: the Roland-Morris Disability Questionnaire (RMDQ) and the Oswestry Disability Index (ODI). In addition, depending on data availability and input from our Advisory Council we will create at least two other crosswalks/links between the PROMIS-29 and other legacy measures for CLBP (e.g., the Back Pain Functional Scale) or legacy measures for other types of chronic pain (e.g., the Neck Disability Index for chronic neck pain).

To address the second challenge, in Aim 2 we will evaluate and refine the chronic pain impact stratification scheme proposed by the NIH Research Task Force on chronic low back pain. The proposed scheme uses the Impact Stratification Score (ISS) which is calculated using 9 items from the PROMIS-29. This ISS was intended to identify and categorize patients with chronic pain into groups based on the severity of their condition so that treatment can be better targeted. We will first evaluate the ISS and its properties to determine whether they are stable across different samples and determine whether they can be improved. After we have finalized the components and calculation of the ISS, we will examine its effect on the impacts of chronic pain (e.g., health-related quality of life, healthcare utilization, worker productivity) to identify meaningful cut-points to use to stratify chronic pain patients into subgroups who exhibit different levels of chronic pain impact.

Three types of data will be used in the analyses to address Aims 1 and 2: data from existing datasets built during other studies, data collected from an anonymous national convenience sample using Amazon's Mechanical Turk (MTurk) crowdsourcing platform, and data from members of the probability-based nationally representative KnowledgePanel. Aim 3 will evaluate whether MTurk is a reliable, efficient method to collect data on individuals with chronic pain. One part of this evaluation will involve comparison of the results from MTurk to what was found using KnowledgePanel.

ELIGIBILITY:
Inclusion Criteria:

* adult
* self-described chronic pain
* member of one of the panels (MTurk or KnowledgePanel) we are using for data collection

Exclusion Criteria:

* unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We have two cohorts. Both will have similar inclusion and exclusion criteria. The first from MTurk is a non-probability sample, and the second is from KnowledgePanel and is a probability-based sample, but one that has been established by the group who owns this panel.
Sampling Method: Non-Probability Sample
Enrollment: 11146 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-10-02 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline only
  Measure of function for those with chronic back pain; range 0-100; higher is worse
Roland-Morris Disability Questionnaire (RMDQ) | Baseline only
  Measure of function for those with chronic back pain; range 0-100; higher is worse
Impact Stratification Score (ISS) | Baseline only
  Measure of the level of impact chronic pain has on individual's lives; range 8-50; higher is worse

SECONDARY OUTCOMES:
PROMIS pain intensity | Baseline only
  Measure of pain intensity; range 0-10; higher is worse
PROMIS pain interference | Baseline only
  Measure of the amount of interference pain causes in life; range 4-20; higher is worse
PROMIS physical function | Baseline only
  Measure of the impact of a condition on physical function; range 4-20; higher is worse
Change in Impact Stratification Score (ISS) | Baseline and 3 months
  Measure of the change in the level of impact chronic pain has on individual's lives; range -42 to +42; positive values are a worsening of impact

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M Herman, ND, PhD, Principal Investigator — RAND
Locations (1):
- Online recruitment only - nationwide, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All data collected is shared.
Supporting Information: Study Protocol
Time Frame: Data were made available 3/8/24
Access Criteria: All researchers with access to ICPSR - openicpsr-198049
URL: https://www.icpsr.umich.edu/

REFERENCES:
- [Result] Edelen MO, Rodriguez A, Herman P, Hays RD. Crosswalking the Patient-Reported Outcomes Measurement Information System Physical Function, Pain Interference, and Pain Intensity Scores to the Roland-Morris Disability Questionnaire and the Oswestry Disability Index. Arch Phys Med Rehabil. 2021 Jul;102(7):1317-1323. doi: 10.1016/j.apmr.2021.02.014. Epub 2021 Mar 5. PMID 33684368
- [Result] Herman PM, Edelen MO, Rodriguez A, Hilton LG, Hays RD. A protocol for chronic pain outcome measurement enhancement by linking PROMIS-29 scale to legacy measures and improving chronic pain stratification. BMC Musculoskelet Disord. 2020 Oct 10;21(1):671. doi: 10.1186/s12891-020-03696-2. PMID 33038933
- [Result] Dunbar MS, Rodriguez A, Edelen MO, Hays RD, Coulter ID, Siconolfi D, Herman PM. Longitudinal Associations of PROMIS-29 Anxiety and Depression Symptoms With Low Back Pain Impact in a Sample of U.S. Military Service Members. Mil Med. 2023 Mar 20;188(3-4):e630-e636. doi: 10.1093/milmed/usab339. PMID 34417805
- [Result] PROMIS(R) Health Organization (PHO) 2021 Conference Abstracts. J Patient Rep Outcomes. 2021 Oct 1;5(Suppl 1):90. doi: 10.1186/s41687-021-00349-3. No abstract available. PMID 34595566
- [Result] Hays RD, Orlando Edelen M, Rodriguez A, Herman P. Support for the Reliability and Validity of the National Institutes of Health Impact Stratification Score in a Sample of Active-Duty U.S. Military Personnel with Low Back Pain. Pain Med. 2021 Oct 8;22(10):2185-2190. doi: 10.1093/pm/pnab175. PMID 34022052
- [Result] Hays RD, Shannon ZK, Long CR, Spritzer KL, Vining RD, Coulter ID, Pohlman KA, Walter JA, Goertz CM. Health-Related Quality of Life Among United States Service Members with Low Back Pain Receiving Usual Care Plus Chiropractic Care vs Usual Care Alone: Secondary Outcomes of a Pragmatic Clinical Trial. Pain Med. 2022 Aug 31;23(9):1550-1559. doi: 10.1093/pm/pnac009. PMID 35060609
- [Result] Hilton LG, Coulter ID, Ryan GW, Hays RD. Comparing the Recruitment of Research Participants With Chronic Low Back Pain Using Amazon Mechanical Turk With the Recruitment of Patients From Chiropractic Clinics: A Quasi-Experimental Study. J Manipulative Physiol Ther. 2021 Oct;44(8):601-611. doi: 10.1016/j.jmpt.2022.02.004. Epub 2022 Jun 18. PMID 35728997
- [Result] Hays RD, Slaughter ME, Spritzer KL, Herman PM. Assessing the Significance of Individual Change in 2 Samples of Patients in Treatment for Low Back Pain Using 5 Different Statistical Indicators. J Manipulative Physiol Ther. 2021 Nov-Dec;44(9):699-706. doi: 10.1016/j.jmpt.2022.03.002. Epub 2022 Jun 23. PMID 35753878
- [Result] Herman PM, Coulter ID, Hays RD, Rodriguez A, Edelen MO. A Scoping Review of Chronic Low Back Pain Classification Schemes Based on Patient-Reported Outcomes. Pain Physician. 2022 Sep;25(6):471-482. PMID 36122256
- [Result] Hays RD, Slaughter M, Rodriguez A, Edelen MO, Herman PM. Analyses of Cross-Sectional Data to Link the PEG With the Patient Reported Outcomes Measurement and Information System (PROMIS) Global Physical Health Scale. J Pain. 2022 Nov;23(11):1904-1911. doi: 10.1016/j.jpain.2022.06.006. Epub 2022 Jun 26. PMID 35768043
- [Result] Hays RD, Qureshi N, Edelen M, Rodriguez A, Slaughter M, Herman PM. Crosswalking the National Institutes of Health Impact Stratification Score to the PEG. Arch Phys Med Rehabil. 2023 Mar;104(3):425-429. doi: 10.1016/j.apmr.2022.08.006. Epub 2022 Aug 27. PMID 36030893
- [Result] Qureshi N, Edelen M, Hilton L, Rodriguez A, Hays RD, Herman PM. Comparing Data Collected on Amazon's Mechanical Turk to National Surveys. Am J Health Behav. 2022 Oct 17;46(5):497-502. doi: 10.5993/AJHB.46.5.1. PMID 36333833
- [Result] Rodriguez A, Edelen MO, Herman PM, Hays RD. Unpacking the impact of chronic pain as measured by the impact stratification score. BMC Musculoskelet Disord. 2022 Sep 23;23(1):884. doi: 10.1186/s12891-022-05834-4. PMID 36151555
- [Result] Herman PM, Qureshi N, Arick SD, Edelen MO, Hays RD, Rodriguez A, Weir RL, Coulter ID. Definitions of Chronic Low Back Pain From a Scoping Review, and Analyses of Narratives and Self-Reported Health of Adults With Low Back Pain. J Pain. 2023 Mar;24(3):403-412. doi: 10.1016/j.jpain.2022.10.012. Epub 2022 Oct 23. PMID 36283654